CLINICAL TRIAL: NCT07311213
Title: EXPLORATIONS CELLULAIRES - CELLULES PLURIPOTENTES INDUITES DES SUJETS PRESENTANT UN TSA, DE LEURS APPARENTES, ET DE TEMOINS
Brief Title: GENES AND AUTISM - IPSC
Acronym: IPSC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: APHP (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C22-14
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Autism Disorder; ASD
Keywords: Autism, Genes, Phenotype, Complex Heritability
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probands with Autism Spectrum Disorder, (N=200). (Other): All subjects included in this study will be drawn from the population of subjects already included in the studies entitled 'Genes and Autism' promoted by Inserm (NCT02628808/C07-33 and NCT04727489/C16-89).
  Patients are diagnosis ASD according to DSM-V criteria and carry genetic variations known to be associated with autism (whether rare or common).
  Interventions: Other: Blood Sample : isolation of peripheral blood mononuclear cells (PBMCs)
- Controls without Autism Spectrum Disorder (Other): At least, 24 months old (N=150) All subjects included in this study will be drawn from the population of subjects already included in the studies entitled 'Genes and Autism' promoted by Inserm (NCT02628808/C07-33 and NCT04727489/C16-89).
  Interventions: Other: Blood Sample : isolation of peripheral blood mononuclear cells (PBMCs)
- Relatives of the probands with ASD (Other): Adult relatives of controls with ASD (N=100) All subjects included in this study will be drawn from the population of subjects already included in the studies entitled 'Genes and Autism' promoted by Inserm (NCT02628808/C07-33 and NCT04727489/C16-89).
  Interventions: Other: Blood Sample : isolation of peripheral blood mononuclear cells (PBMCs)

INTERVENTIONS:
Other: Blood Sample : isolation of peripheral blood mononuclear cells (PBMCs) — Participation in this study requires a single visit per participant. This study only requires a blood sample (5 to 30 minutes) to be taken at the CIC at Robert-Debré Hospital, Paris 19th arrondissement.
  This blood sample will enable the isolation of peripheral blood mononuclear cells (PBMCs). HIV, HCV and HBV serology will also be performed.

SUMMARY:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder characterized by deficits in social interaction and verbal and non-verbal communication (DSM-5, 2013), affecting approximately 2% of the general population. In 5 to 40% of cases, genetic factors are identified as the cause of these disorders, with prevalence depending on the technique used (exomes and/or SNP arrays) and the associated intellectual deficit. In the majority of cases, the aetiology remains unknown. Studies of microdeletions/microduplications (copy number variants) or Whole Exome Sequencing and Whole Genome Sequencing (Single Nucleotide Variants) show the involvement of numerous genes in the predisposition to autism. ASD remains a genetically heterogeneous disorder, as more than 250 genes have been associated with ASD to date.

The main objective of the project is to continue identifying genetic factors, and also to understand the biological mechanisms involved in the emergence of autistic symptoms.

Identifying biological pathways is an essential step in developing new therapeutic strategies. In addition, one of the major challenges of this study is to better understand the phenotype/genotype relationships in ASD. This requires in-depth knowledge of the phenotypic characteristics of ASD participants and their families, as well as neurotypical populations. This study combines the scientific expertise of researchers specializing in molecular biology, phenotypic exploration (clinical, cognitive, MRI, EEG, biochemistry, immunology), and the use of pre-therapeutic cellular models (iPSCs, neural precursors, organoids).

The objectif of this work is the identification of numerous genes associated with ASD and involved in synaptic formation and regulation: NLGN3-4, SHANK1 and SHANK3, CNTN-6, and CNTNAP4. This work was combined with in-depth phenotypic explorations of ASD participants and their relatives. It has made it possible to clarify the neuroanatomical characteristics of ASD participants and their genetic substrate, as well as the underlying cognitive processes.

All of this work opens up new prospects for identifying new therapeutic targets using preclinical cell models (IPS, neural progenitors, organoids) developed in particular by I-Stem and Human Technopole.

DETAILED DESCRIPTION:
* Aim 1 : To clarify the biological mechanisms associated with genetic variations identified in participants with ASD by studying dedifferentiated cells transformed into induced neurons or organoids. This objective will be achieved using a population of individuals with ASD, a population of relatives and a population of controls.
* Aim 2 : To study the cellular mechanisms affected by the presence of abnormalities identified in participants with ASD. The use of pluripotent cells derived into neurons or organoids is a major tool for understanding the pathophysiology of cell development and pathways in autism. These derived neurons are an indispensable proxy for the biological understanding of ASD.
* Aim 3 : To identify new therapeutic approaches , by using pluripotent cells and organoids to perform high-throughput screening of pharmacological compounds.

ELIGIBILITY:
Inclusion Criteria:

● For all participants :

* 1) Be Included in the "Genes and Autism" protocol (C07-33 or C16-89).
* 2) Affiliated to the social insurance, Universal Health Coverage or any equivalent system.

  →As a Reminder : C07-33 inclusion criteria

  ● Participants with ASD.
* 1) Autistic patients must meet the diagnostic criteria of DSM-IV [American Psychiatric Association, 1994] and the criteria of ADI-R (Autism Diagnostic Interview-Revised, Lord et al., 1994) and ADOS for autism.

..Or.. Patients with Asperger's syndrome must meet the DSM-IV criteria as well as the ASDI criteria for Asperger's syndrome (Asperger Syndrome Diagnostic Interview, Gillberg et al., 2001) and the ADOS for autism spectrum disorders.

..Or.. Patients with ASD must meet diagnostic criteria of DSM-IV and ADOS criteria for autism spectrum disorders

* 2) Be at least 2 years old, with no upper age limit
* 3) Somatic state compatible with blood test

  ● Adult controls and adult relatives of controls
* 1) Be between 18 and 65 years old
* 2) Somatic and intellectual state compatible with blood test

  ● Controls with mental retardation
* 1) Minimum age of 2 yearsIQ < 70Child controls
* 2) Minimum age of 2 years

  →As a Reminder : inclusion criteria C16-89

  ● Probands with ASD
* 1) Meet the diagnostic criteria for ASD of the of DSM-5 [American Psychiatric Association, 2012]. The diagnosis will be based on a consensus between the clinical expertise of expert clinicians, the scores of the Autism Diagnostic Interview-Revised (ADI-R) (Lord et al, 2003) and those of the Autism Diagnosis Observational Scale (ADOS-2) (Lord et al, 1994)
* 2) Be at least 24 months old with no upper age limit
* 3) Somatic state compatible with a blood test
* 4) Affiliation to the Social Insurance
* 5) Signature of informed consent by the applicant or by the holders of parental authority if the subject is a minor or by the guardian if the subject is under guardianship

  ● Controls wihout ASD
* 1) At least 24 months old
* 2) Somatic and Intellectual state compatible with a blood test
* 3) Affiliation in the Social Insurance
* 4) Signature of informed consent by the subject or by holders of parental authority if the subject is a minor, or by the guardian if the subject is under guardianship

  ● Relatives of the probands with ASD or of controls without ASD
* 1) At least 24 months old
* 2) Somatic and intellectual state compatible with blood test
* 3) Affiliation to the Social Insurance
* 4) Signature of informed consent by the subject or by the holders of parental authority if the subject is a minor or by the guardian if the subject is under guardianship

Exclusion Criteria:

* For all participants

  * 1) Refusal to have a blood test
  * 2) Medical illness (including psychiatric disorder) not yet fully stabilised and making participation in the study impossible
  * 3) Person subject to a mesure of lagal protection
  * 4) Known serology : VIH+ or VBH+ or VCH+

    * As a reminder : exclusion criteria C07-33
  * 1) For all participants : Severe Intelectual Deficiency (IQ,35 or developmental age <18 months)
  * 2) Controls : Neurological or psychiatric history other than mental retardation

    o Psychiatric history, except for mental retardation, assessed using the DIGS (Diagnostic Interview for Genetic Studies, Nurnberger et al., 1994) for adults or the Kiddie-SADS (Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children, Orvaschel et al., 1982)

    o History of epileptic episodes

    o Immunosuppressive treatment or known immunoinflammatory disease

    →As a reminder : exclusion criteria C16-89
  * 1) Probands with Autism Spectrum Disorder

    o Severe intellectual disability (IQ<35 or developmental age <18 months)
  * 2) Controls (neurotypical development)

    o Identified intellectual disorder or cognitive developmental disorder
    * Personal psychiatric history of schizophrenia, bipolar disorder, substance use disorders (except tobacco), recurrent depression (>2 episodes, lifetime), severe unstabilized anxiety disorder
    * History of epilepsy episodes or severe neurological disease
  * 3) Relatives of the TSA applicants or controls

    * Medical condition (psychiatric or somatic) not compatible with inclusion

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2041-02-01 (Estimated); Study Completion 2041-02-01 (Estimated)

PRIMARY OUTCOMES:
Isolation of peripheral blood mononuclear cells (PBMCs) | Inclusion visit
  Blood sample to be taken from individuals with ASD, a population of relatives, and a population of controls.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pr Bourgeron, Professor, Study Director — Institut Pasteur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.fondation-fondamental.org/faire-avancer-la-recherche/les-projets-de-fondamental/projet-genes-et-autisme